CLINICAL TRIAL: NCT06248476
Title: Effect of Intermittent Theta Burst Stimulation and Repetitive Transcranial Magnetic Stimulation Combined With Robotic Rehabilitation on Ambulation and Lower Extremity Motor Function in Chronic Spinal Cord Injury Patients
Brief Title: Intermittent Theta Burst Stimulation and Repetitive Transcranial Magnetic Stimulation Combined With Robotic Rehabilitation on Ambulation in Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Naz Kalem, Asist. Dr., Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-5440
Record Dates: First submitted 2024-01-25; First posted 2024-02-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injury; rTMS; iTBS; Ambulation; Lower extremity motor function
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- iTBS + robotic rehabilitation (Active Comparator): iTBS combined with robotic rehabilitation and conservative treatment applied to patients with chronic incomplete spinal cord injury
  Interventions: Device: Transcranial Magnetic Stimulation
- rTMS + robotic rehabilitation (Active Comparator): rTMS combined with robotic rehabilitation and conservative treatment applied to patients with chronic incomplete spinal cord injury
  Interventions: Device: Transcranial Magnetic Stimulation
- sham iTBS + robotic rehabilitation (Sham Comparator): Sham iTBS combined with robotic rehabilitation and conservative treatment applied to patients with chronic incomplete spinal cord injury
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation is non-invasive stimulation technique which modifies cortical excitability through forming magnetic field

SUMMARY:
Comparison of different types of transcranial magnetic stimulation techniques which are intermittent theta burst stimulation (iTBS) and high frequency repetitive transcranial magnetic stimulation (rTMS) in patients with spinal cord injury

DETAILED DESCRIPTION:
iTBS lasts shorter than rTMS so that this technique comfortable than rTMS for both patients and also physicians. Aim of this study is to compare effectiveness of this techniques. If results are same, iTBS can be used instead of rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete spinal cord injury (ASIA C and D)
* 12 months after spinal cord injury
* At least 10 meters walking independent or with canadian, walker or walking stick
* Put signature to approved form

Exclusion Criteria:

* Epileptic seizure
* Pacemaker
* Pregnancy
* Neurological disease different from spinal cord injury
* Metalic implant in brain or scalp
* Brain surgery
* Orthopedic problem in lower extremity
* Malignity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Lower extremity motor score | Before treatment (0. week), finishing time of treatment (2.week), 4 weeks after finishing time of treatment (6.week)
  Assesment of lower extremity key motor muscle function according to American Spinal Injury Association

SECONDARY OUTCOMES:
Walking index for spinal cord injury II | Before treatment (0. week), finishing time of treatment (2.week), 4 weeks after finishing time of treatment (6.week)
  Assesment of ambulation ability after spinal cord injury
Spinal cord injury independence measurement III (SCIM III) | Before treatment (0. week), finishing time of treatment (2.week), 4 weeks after finishing time of treatment (6.week)
  Assesment of independence of daily living activities in patients with spinal cord injury
10 meter walking test | Before treatment (0. week), finishing time of treatment (2.week), 4 weeks after finishing time of treatment (6.week)
  Patients with spinal cord injury walk between two markers, that distance is 10 meters
Time up and go test | Before treatment (0. week), finishing time of treatment (2.week), 4 weeks after finishing time of treatment (6.week)
  Patients sit chair, then walk 3 meter, return and sit again
Motor evoked potential | Before treatment (0. week), finishing time of treatment (2.week), 4 weeks after finishing time of treatment (6.week)
  For assesment of cortical excitability

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Training and Research Hospital, Ankara, Çankaya, Turkey (Türkiye)